CLINICAL TRIAL: NCT06825312
Title: Immunogenicity, Safety, and Antibody Persistence of Different Immunization Strategies Against Japanese Encephalitis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Liaoning Chengda Biotechnology CO., LTD (Industry)
Collaborators: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDB-JE-PM-2023002
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Japanese Encephalitis Vaccine
MeSH Terms: interventions — Japanese Encephalitis Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1 (4 doses of JEV-I) (Experimental): Participants will receive 2 doses of JEV-I (7-10 days apart) at 8 months of age, 1 dose of JEV-I at 24 months of age, and 1 dose of JEV-I at 6 years of age.
  Interventions: Biological: Japanese Encephalitis Vaccine (Vero Cell), Inactivated
- Group 2 (4 doses of JEV-I) (Experimental): Participants will receive 2 doses of JEV-I (28-35 days apart) at 8 months of age, 1 dose of JEV-I at 24 months of age, and 1 dose of JEV-I at 6 years of age.
  Interventions: Biological: Japanese Encephalitis Vaccine (Vero Cell), Inactivated
- Group 3 (2 doses of JEV-I and 1 dose of JEV-L) (Experimental): Participants will receive 2 doses of JEV-I (7-10 days apart) at 8 months of age and 1 dose of JEV-L at 24 months of age.
  Interventions: Biological: Japanese Encephalitis Vaccine (Vero Cell), Inactivated; Biological: Japanese Encephalitis Vaccine, Live
- Group 4 (1 dose of JEV-L and 2 doses of JEV-I) (Experimental): Participants will receive 1 dose of JEV-L at 8 months of age and 2 doses of JEV-I (7-10 days apart) at 24 months of age.
  Interventions: Biological: Japanese Encephalitis Vaccine (Vero Cell), Inactivated; Biological: Japanese Encephalitis Vaccine, Live
- Group 5 (1 dose of JEV-L and 2 doses of JEV-I) (Experimental): Participants will receive 1 dose of JEV-L at 8 months of age, 1 dose of JEV-I at 24 months of age, and 1 dose of JEV-I at 6 years of age.
  Interventions: Biological: Japanese Encephalitis Vaccine (Vero Cell), Inactivated; Biological: Japanese Encephalitis Vaccine, Live
- Group 6 (2 doses of JEV-L) (Active Comparator): Participants will receive 2 doses of JEV-L at 8 months of age, and 1 dose of JEV-L at 24 months of age.
  Interventions: Biological: Japanese Encephalitis Vaccine, Live

INTERVENTIONS:
Biological: Japanese Encephalitis Vaccine (Vero Cell), Inactivated — 0.5ml for each dose, manufactured by Liaoning Chengda Biotechnology Co., Ltd., administered in the deltoid area of lateral arm by intramuscular injection.
  Arms: Group 1 (4 doses of JEV-I); Group 2 (4 doses of JEV-I); Group 3 (2 doses of JEV-I and 1 dose of JEV-L); Group 4 (1 dose of JEV-L and 2 doses of JEV-I); Group 5 (1 dose of JEV-L and 2 doses of JEV-I)
Biological: Japanese Encephalitis Vaccine, Live — 0.5ml for each dose, manufactured by Chengdu Institute of Biological Products Co., Ltd., administered subcutaneously in the lower part of the deltoid area of lateral arm.
  Arms: Group 3 (2 doses of JEV-I and 1 dose of JEV-L); Group 4 (1 dose of JEV-L and 2 doses of JEV-I); Group 5 (1 dose of JEV-L and 2 doses of JEV-I); Group 6 (2 doses of JEV-L)

SUMMARY:
The main objective of this study is to evaluate the persistence of Japanese encephalitis antibodies in participants at the age of 6, after they have followed different Japanese encephalitis vaccination schedules. Furthermore, the study will assess the immunogenicity and antibody persistence of primary immunization across different Japanese encephalitis vaccination schedules, as well as the immunogenicity following booster immunizations within these schedules. The safety of each vaccine dose will also be evaluated.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, non-inferiority study. Healthy children aged 8 months will be invited to participate and randomly allocated to six groups (Group 1 to Group 6) in a 1:1:1:1:1:1 ratio. They will be administered the inactivated Japanese encephalitis vaccine (JEV-I) and/or the live attenuated Japanese encephalitis vaccine (JEV-L) based on the six schedules delineated in the protocol. The primary immunization will be administered to participants at 8 months of age, and a booster dose will be given at 24 months of age. Additionally, participants in Groups 1, 2, and 5 will receive an additional booster dose at the age of 6.

Blood samples (3 mL) will be collected from participants at 8 months, 24 months, and 6 years of age. Samples will be taken before vaccination and 30 days after it for detecting Japanese encephalitis neutralizing antibodies. The titers of these antibodies will be assayed via the 50% plaque reduction neutralization test. Those in groups 3, 4, and 6 who've completed all immunization procedures by 24 months old will have a blood sample taken at 6 years old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 8 months who are permanent residents of the study area.
* Legal guardians can understand the requirements and processes of the study, provide written informed consent, and comply with all procedures as required by the clinical research protocol.
* Able to receive the full course of Japanese encephalitis vaccinations according to the immunization strategy in the research protocol, including receiving the primary immunization at 8 months of age and the booster immunizations at 24 months of age and 6 years of age.

Exclusion Criteria:

* Unable to finish the full course of primary and booster immunizations at the study area, and unable to fulfill the follow-up visits prescribed in the protocol.
* Non-compliance with the vaccination strategy for each group, as stated in the protocol, regarding Japanese encephalitis vaccines with proper doses and varieties.
* Allergic to any component of the study vaccine or having a history of allergic reactions to any vaccines.
* Having a history of symptoms or signs of neurological diseases or other contraindications for Japanese encephalitis vaccine vaccination.
* Having used immunosuppressants or blood products following birth.
* Receiving other vaccines simultaneously while receiving the Japanese encephalitis vaccine of this project.
* Any conditions that may interfere with the evaluation of the study, as deemed by the researcher.

Ages: 8 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Testing Seropositive for Japanese Encephalitis Neutralizing Antibodies | 4 years after the booster vaccination at 24 months of age
  The persistence of immunity following various Japanese encephalitis (JE) vaccination schedules is evaluated based on the proportion of participants exhibiting seropositivity for JE neutralizing antibodies at 6 years of age. Seropositivity is defined as a JE neutralizing antibody titer of at least 1:10, as ascertained by the 50% plaque reduction neutralization test.

SECONDARY OUTCOMES:
Seroconversion Rates of Japanese Encephalitis Neutralizing Antibodies after Primary vaccination | 30 days post-primary immunization
  The seroconversion rate is defined as the percentage of participants with a change in Japanese Encephalitis neutralizing antibody titer from <1:10 at baseline (pre-vaccination) to a titer of ≥1:10 30 days post-vaccination, or a 4-fold or greater rise from the baseline, as measured by the 50% plaque reduction neutralization test
Geometric Mean Titer of Japanese Encephalitis Neutralizing Antibodies before and after Primary Immunization | pre-primary immunization (Day 0) and 30 days post-primary immunization
Percentage of Participants Testing Seropositive for Japanese Encephalitis Neutralizing Antibodies before and after Primary Immunization | pre-primary immunization (Day 0) and 30 days post-primary immunization
  Seropositivity is defined as a Japanese Encephalitis neutralizing antibody titer of at least 1:10, as ascertained by the 50% plaque reduction neutralization test.
Seroconversion Rates of Japanese Encephalitis Neutralizing Antibodies after Booster vaccination | 30 days post-booster immunization
  The seroconversion rate is defined as the percentage of participants with a change in Japanese Encephalitis neutralizing antibody titer from <1:10 at baseline (pre-vaccination) to a titer of ≥1:10 30 days post-vaccination, or a 4-fold or greater rise from the baseline, as measured by the 50% plaque reduction neutralization test
Geometric Mean Titer of Japanese Encephalitis Neutralizing Antibodies before and after booster Immunization | pre-booster immunization (Day 0) and 30 days post-booster immunization
Percentage of Participants Testing Seropositive for Japanese Encephalitis Neutralizing Antibodies before and after booster Immunization | pre-booster immunization (Day 0) and 30 days post-booster immunization
  Seropositivity is defined as a Japanese Encephalitis neutralizing antibody titer of at least 1:10, as ascertained by the 50% plaque reduction neutralization test.
Incidence of any Local and Systemic Adverse Events Within 30 Days of Each Vaccination | within 30 days of each vaccination
  Adverse events will be collected through a combination of proactive visits by researchers and participant reports

CONTACTS AND LOCATIONS:
Overall Officials: Huanyu Wang, Study Director — Liaoning Chengda Biotechnology CO., LTD
Locations (6):
- China (6):
  - Jiashan County Center for Disease Control and Prevention, Jiaxing, Zhejiang
  - Pinghu Center For Disease Control and Prevention, Jiaxing, Zhejiang
  - Dongyang Center for Disease Control and Prevention, Jinhua, Zhejiang
  - Yongkang Center for Disease Control and Prevention, Jinhua, Zhejiang
  - Yuyao Center for Disease Control and Prevention, Ningbo, Zhejiang
  - Jiangshan Center For Disease Control and Prevention, Quzhou, Zhejiang